CLINICAL TRIAL: NCT02168101
Title: Open-Label Study to Determine the Feasibility of MLN9708 as Maintenance After Allogeneic Stem Cell Transplant for Multiple Myeloma, Followed by an Expansion Phase at the Maximum-Tolerated Dose (MTD) - A Phase II Study
Brief Title: Determining the Feasibility of MLN9708 as Maintenance After Allogeneic Stem Cell Transplant for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI MM 42
Record Dates: First submitted 2014-06-12; First posted 2014-06-20 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Multiple Myeloma
Keywords: MLN9708; allogeneic stem cell transplant; multiple myeloma; ixazomib; autologous stem cell transplant
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MLN9708 - 2.3 mg (Experimental): Patients will be enrolled between Days 45 and 120 after allogeneic transplant and will receive a weekly dose of 2.3 mg of MLN9708 on Days 1, 8, and 15 of each 28-day cycle for 6 cycles.
  Interventions: Drug: MLN9708
- MLN9708 - 3 mg (Experimental): Patients will be enrolled between Days 45 and 120 after allogeneic transplant and will receive a weekly dose of 3 mg of MLN9708 on Days 1, 8, and 15 of each 28-day cycle for 6 cycles.
  Interventions: Drug: MLN9708
- MLN9708 - 4 mg (Experimental): Patients will be enrolled between Days 45 and 120 after allogeneic transplant and will receive a weekly dose of 4 mg of MLN9708 on Days 1, 8, and 15 of each 28-day cycle for 6 cycles.
  Interventions: Drug: MLN9708

INTERVENTIONS:
Drug: MLN9708 — Patients will be enrolled between Days 45 and 120 after allogeneic transplant and will receive MLN9708 orally (PO) as monotherapy on Days 1, 8, and 15 of each 28-day cycle for 6 cycles. Up to 18 patients will be enrolled in a dose-escalation phase to determine the maximum tolerated dose (MTD).
  Dose-Escalation Phase: MLN9708 will be administered orally (PO) as monotherapy. Dosing will start at 2.3 mg. If acceptable tolerability is demonstrated, escalations will be made to 3 mg and to a maximum-planned dose (MPD) of 4 mg.
  Other Names: ixazomib

SUMMARY:
The purpose of the study is to determine the safety of MLN9708 as maintenance therapy following allogeneic stem cell transplant in patients with multiple myeloma.

DETAILED DESCRIPTION:
Although multiple myeloma is considered fatal, survival has dramatically improved over the last two decades with the introduction of more effective treatment options. Proteasome inhibitors have an anti-myeloma effect and are often used as either initial treatment or at relapse in patients with multiple myeloma. MLN9708 is an orally bioavailable, potent, reversible inhibitor of the 20S proteasome. Phase I studies have shown MLN9708 to be very well tolerated with minimal peripheral neuropathy. It has also shown impressive anti-myeloma activity in both the relapsed/refractory setting and the upfront setting (Kumar et al. 2011, Berdeja et al. 2011, Richardson et al. 2011). These characteristics make MLN9708 an ideal proteasome inhibitor to use after allogeneic stem cell transplant. In this Phase II, open-label, multicenter, non-randomized study the investigators will investigate the role of MLN9708 as maintenance after allogeneic stem cell transplant in patients with high-risk multiple myeloma, and in patients with multiple myeloma who have relapsed after an autologous stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

KEY POINTS:

1. Symptomatic multiple myeloma or asymptomatic myeloma with myeloma-related organ damage diagnosed according to standard criteria in patients who received allogeneic transplant due to high-risk prognostic features, such as, but not limited to:

   * Chromosome 17p, partial deletion [del(17p)], t(4;14), t(14;16), t(14;20)
   * Plasma cell leukemia
   * PFS of less than 2 years after autologous stem cell transplant
2. Evidence of engraftment of neutrophils (absolute neutrophil count [ANC] >1000 cells/mm3) and platelets (platelets >60,000 cells/mm3) [dose escalation phase] and >50,000 cells/mm3 [dose expansion phase]).
3. Achievement of at least a PR prior to allogeneic stem cell transplant
4. Adequate liver and kidney function
5. Ability to swallow oral medication
6. Absence of gastrointestinal symptoms that precludes oral intake and absorption of MLN9708
7. Off antibiotics and amphotericin B formulations, voriconazole or other anti-fungal therapy for the treatment of proven, probable or possible infections
8. ECOG of ≤ 2
9. Life expectancy ≥3 months
10. Ability to understand the nature of this study and give written informed consent

Exclusion Criteria:

1. Patients with progressive disease when compared to pre-transplant staging as defined by IMWG Uniform Response criteria for Multiple Myeloma.
2. Umbilical cord blood transplant
3. Patients with > Grade 2 peripheral neuropathy with pain, or ≥ Grade 3 peripheral neuropathy per NCI CTCAE Version 4.0
4. Patients with uncontrolled bacterial, viral, or fungal infections
5. New York Heart Association (NYHA) Class III or IV heart failure uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
6. Patients who are pregnant or breastfeeding
7. Most recent chemotherapy ≤21 days and ≤ Grade 1 chemotherapy-related side effects, with the exception of alopecia
8. Use of a study drug ≤21 days or 5 half-lives (whichever is shorter) prior to the first dose of MLN9708. For study drugs for which 5 half-lives is ≤21 days, a minimum of 10 days between termination of the study drug and administration of MLN9708 is required.
9. Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤14 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy
10. Major surgical procedures ≤14 days of beginning study drug, or minor surgical procedures ≤7 days. No waiting is required following port-a-cath placement.
11. Ongoing or active systemic infection. Known diagnosis of human immunodeficiency virus, hepatitis B, or hepatitis C
12. Central Nervous System involvement
13. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
14. Systemic treatment with moderate and strong inhibitors of cytochrome P450 (CYP) 1A2, CYP3A, or clinically significant CYP3A inducers, or use of Ginkgo biloba or St. John's wort within 14 days before study drug administration in the study.
15. Presence of other active cancers, or history of treatment for invasive cancer ≤5 years. Patients with Stage I cancer who have received definitive local treatment and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e., non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
16. Graft versus host disease > Grade 2; or GVHD grade 1 or Grade 2 which requires > 0.5 mg/kg methylprednisolone, or equivalent.

There are additional Inclusion/Exclusion criteria. The Study Center will determine if you meet all criteria and will answer any questions you may have about the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-09; Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Bachier, MD, Study Chair — Texas Transplant Institute
Locations (4):
- United States (4):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Oncology Hematology Care, Cincinnati, Ohio
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Texas Transplant Institute, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- MLN9708 - 2.3 mg: Patients will be enrolled between Days 45 and 120 after allogeneic transplant and will receive a weekly dose of 2.3 mg of MLN9708 orally (PO) on Days 1, 8, and 15 of each 28-day cycle for 6 cycles.
Period: Overall Study
Arm/Group | MLN9708 - 2.3 mg | MLN9708 - 3 mg | MLN9708 - 4 mg
Started | 3 | 3 | 3
Completed | 1 | 1 | 2
Not Completed | 2 | 2 | 1
Not completed — Death | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of MLN9708.
Groups:
- Total: Total of all reporting groups
Arm/Group | MLN9708 - 2.3 mg | MLN9708 - 3 mg | MLN9708 - 4 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Continuous [Median (Full Range); unit: years] | 57 [49 to 64] | 47 [45 to 61] | 44 [27 to 44] | 47 [27 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 6
  Male | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 3 | 3 | 2 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Phase I Patients Receiving 2.3mg, 3mg, or 4mg MLN9708 Experiencing a Dose-Limiting Toxicity (DLT) to Determine the Maximum Tolerated Dose
Description: The maximum tolerated dose (MTD) of MLN9708 will be determined as the dose at which ≤1 of 6 patients experiences a DLT during one cycle (28 days) of therapy utilizing the National Cancer Institute Common Technology Criteria for Adverse Events (NCI CTCAE) v4.0
Time Frame: Collected from day of first dose to the end of the first treatment cycle, up to 28 days
Population: All patients who received at least one dose of MLN9708.
Measure: Count of Participants; unit: Participants
Arm/Group | MLN9708 - 2.3 mg | MLN9708 - 3 mg | MLN9708 - 4 mg
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Grade 3/4/5 Serious Adverse Events and Adverse Events as a Measure of Safety of MLN9708 When Used as Maintenance After Allogeneic Stem Cell Transplant for Multiple Myeloma Multiple Myeloma
Description: Defined as the number of participants with treatment-emergent grade 3/4/5 adverse events/serious adverse events utilizing the National Cancer Institute Common Technology Criteria for Adverse Events (NCI CTCAE) v4.0 determined to be related to MLN9708.
Time Frame: Defined as the time from Day 1 of study drug administration until 30 days after treatment completion for up to 2 years.
Population: All patients who received at least one dose of MLN9708.
Measure: Count of Participants; unit: Participants
Arm/Group | MLN9708 - 2.3 mg | MLN9708 - 3 mg | MLN9708 - 4 mg
Number analyzed (Participants) | 3 | 3 | 3
Participants | 1 | 2 | 2

3. Secondary Outcome: Median Progression-Free Survival (PFS) at 2 Years Post-maintenance Therapy
Description: PFS is measured from the date of first protocol treatment until date of disease progression or death occurs, or date of last adequate tumor assessment using the International Myeloma Working Group Uniform Response Criteria. IMWG disease progression is defined as an increase of ≥ 25% from the nadir in at least one of the following criteria: 1) serum M-protein, 2) urine M-protein, 3) only in patients with non-measurable serum and urine M-protein levels: difference in involved and uninvolved FLC levels, 4) Bone marrow plasma cell percentage (absolute % must be ≥10%). OR Disease progression also could include development of new lytic bone lesions or increase from baseline in size of lytic bone lesion(s); development of new soft tissue plasmacytoma(s) or definite increase from nadir in existing soft tissue plasmacytomas; or development of hypercalcemia
Time Frame: every 8 weeks for approximately 24 weeks then every 3 months thereafter for 2 years
Population: All patients with measurable or evaluable disease at baseline who receive at least 1 dose of MLN9708 and undergo at least one post-baseline disease assessment. Pre-specified in Protocol to calculate PFS for all participants and for all patients receiving the MTD. Because the MTD was not reached, this analysis was only performed on all participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- MLN9708 Combined Dose Escalation: Patients will be enrolled between Days 45 and 120 after allogeneic transplant and will receive a weekly dose of either 2.3, 3, or 4 mg of MLN9708 on Days 1, 8, and 15 of each 28-day cycle for 6 cycles.
Arm/Group | MLN9708 Combined Dose Escalation
Number analyzed (Participants) | 8
months | 6.5 [1.9 to 21.7]

4. Secondary Outcome: Median Overall Survival (OS) at 2 Years Post-allogeneic Stem Cell Transplant (ASCT)
Description: Overall survival is measured as the interval from first study treatment until date of death, or date last known alive.
Time Frame: every 8 weeks for approximately 24 weeks after ASCT, then every 3 months thereafter for 2 years.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MLN9708 Combined Dose Escalation
Number analyzed (Participants) | 8
months | NA [6.1 to NA] — Not reached at this time.

5. Secondary Outcome: Number of Participants With Incidence of Chronic Graft-versus-host Disease (cGVHD) After Receiving Allogeneic Stem Cell Transplant and Maintenance With MLN9708
Description: Incidence of chronic Graft-versus-host disease GVHD was assessed based on the National Institutes of Health Consensus Development Project on Criteria for Clinical trials in Acute and Chronic Graft-versus-host-disease (Filipovich et al. 2005) from date of randomization until date of first documented progression, or date of death from any cause.
Time Frame: from date of enrollment every 28 days, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | MLN9708 - 2.3 mg | MLN9708 - 3 mg | MLN9708 - 4 mg
Number analyzed (Participants) | 3 | 3 | 3
Participants | 2 | 2 | 2

6. Secondary Outcome: Number of Participants With Incidence of Acute Graft-versus-host Disease (aGVHD) After Receiving Allogeneic Stem Cell Transplant and Maintenance With MLN9708
Description: Incidence of acute Graft-versus-host disease GVHD was assessed based on the National Institutes of Health Consensus Development Project on Criteria for Clinical trials in Acute and Chronic Graft-versus-host-disease (Przepiorka et al. 1995) from date of randomization until date of first documented progression, or date of death from any cause.
Time Frame: from date of enrollment every 28 days, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | MLN9708 - 2.3 mg | MLN9708 - 3 mg | MLN9708 - 4 mg
Number analyzed (Participants) | 3 | 3 | 3
Participants | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the start of study treatment, until 30 calendar days after discontinuation or completion of study treatment. All AEs resulting in discontinuation from the study treatment were followed until resolution or stabilization. After 30 days of completion of protocol-specific treatment or discontinuation, only AEs, SAEs, or deaths assessed by the Investigator as treatment related were reported.
Description: Any untoward medical occurrence in a participant regardless of the relationship with the study drug per the Investigator's assessment. Adverse events were evaluated using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0. All-Cause Mortality was assessed in all randomized participants, while Serious and Other (Not Including Serious) Adverse Events was only assessed in participants who received at least one dose of study treatment.
Arm/Group | MLN9708 - 2.3 mg | MLN9708 - 3 mg | MLN9708 - 4 mg
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN9708 - 2.3 mg (N=3) | MLN9708 - 3 mg (N=3) | MLN9708 - 4 mg (N=3)
Pyrexia (General disorders) | 0 | 1 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Graft Versus Host Disease (Immune system disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MLN9708 - 2.3 mg (N=3) | MLN9708 - 3 mg (N=3) | MLN9708 - 4 mg (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypertension (Vascular disorders) | 2 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 2
Dry eye (Eye disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Chills (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0
Temperature intolerance (General disorders) | 1 | 0 | 0
Acute graft versus host disease in skin (Immune system disorders) | 1 | 0 | 0
Chronic graft versus host disease (Immune system disorders) | 1 | 0 | 0
Graft versus host disease (Immune system disorders) | 0 | 1 | 0
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 1
Infected dermal cyst (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood immunoglobulin G decreased (Investigations) | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1
Human metapneumovirus test positive (Investigations) | 0 | 1 | 0
Respiratory syncytial virus test positive (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Bladder discomfort (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-02-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT02168101/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT02168101/SAP_001.pdf